CLINICAL TRIAL: NCT01624402
Title: Ecosystem Focused Therapy in Post Stroke Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH096685 (NIH); R01MH096685 (NIH)
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Depression; Stroke
MeSH Terms: conditions — Depression; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ecosystem Focused Therapy (EFT) (Experimental): Ecosystem Focused Therapy (EFT) follows a structured personalization approach based on the model of adaptive functioning, in which behavior is a function of the person's competence and the demands of the environment.
  Interventions: Behavioral: Ecosystem Focused Therapy (EFT)
- Education on Stroke and Depression (ESD) (Active Comparator): Education on Stroke and Depression (ESD) is home-delivered and imparts education about depression, stroke, and the role of available treatments.
  Interventions: Behavioral: Education on Stroke and Depression (ESD)

INTERVENTIONS:
Behavioral: Education on Stroke and Depression (ESD) — * Each session begins by assessing the subject's and his/her family's level of information in a given area and by identifying misconceptions, thus guiding the selection of educational material.
  * Comprehending illness-related information is a process contaminated by pessimism, denial, misconceptions, and stigma. The role of the ESD therapist is to impart valuable information, despite these complexities.
  * Conveying information is a process. The ESD therapist needs to be aware of where the subject and family are in each session and offer information for which they have readiness to accept.
  * ESD therapists do not engage in additional interventions (e.g., cognitive behavioral therapy, interpersonal therapy, problem solving therapy).
  Arms: Education on Stroke and Depression (ESD)
Behavioral: Ecosystem Focused Therapy (EFT) — 1. EFT offers an action-oriented, new perspective about the subject's recovery;
  2. It provides an adherence enhancement structure;
  3. It offers a problem solving structure to the subject focusing on problems, valued by the subject, and pertinent to daily function;
  4. It helps the family re-engineer its goals, involvement, and plans to accommodate the patient's disability;
  5. It coordinates care with specialized therapists with the goal to increase patient participation in rehabilitation and social activities.
  Arms: Ecosystem Focused Therapy (EFT)

SUMMARY:
Older adults who are stroke survivors can experience many challenges, including depression, cognitive dysfunction, and physical disability. Family members and other caregivers may struggle with helping stroke survivors adjust to life after stroke. This research study involves testing a modified form of problem-solving therapy called Ecosystem Focused Therapy (EFT) to help treat depression in older adult stroke survivors. EFT teaches problem-solving skills to patients to help them cope with problems related to stroke and depression, alters their physical environment to accommodate new needs resulting from stroke, and helps the family or caregiver to assist in the patient's adaptation. In addition this study will compare EFT to an education intervention to see which is more effective in treating depressed stroke survivors.

DETAILED DESCRIPTION:
We propose to study the efficacy of "Ecosystem Focused Therapy" (EFT) in post-stroke depression (PSD), a disorder that afflicts a large number of stroke victims and increases mortality, cognitive impairment, and disability for years after stroke. EFT is a new, home-delivered intervention based on our integrative model of PSD, which originated from our clinical biology and treatment studies in late-life depression. It postulates two main paths to PSD. First, stroke and stroke-repair mechanisms contribute to metabolic changes mediating PSD. Second, a "psychosocial storm" stemming both from the patient's sudden disability and the change in the patient's needs and family life add a biological burden to this cascade of depressogenic events. EFT targets the "psychosocial storm" of PSD and focuses on the reciprocal interaction between the patient's abilities and the challenges of his/her "ecosystem" (family, specialized therapists). EFT follows a structured personalization approach based on the "model of adaptive functioning", in which behavior is a function of the person's competence and the demands of the environment. Thus, EFT continuously "calibrates the environment" to the PSD patient's competence level and targets the PSD "psychosocial storm" through five integrated components: 1) It offers an action-oriented, "new perspective" about the patient's recovery. 2) It provides an "adherence enhancement structure". 3) It offers a "problem solving structure" to the patient focusing on problems, valued by the patient, and pertinent to daily function. 4) It helps the family "reengineer its goals, involvement, and plans" to accommodate the patient's disability. 5) It "coordinates care with specialized therapists" with the goal to increase patient participation in rehabilitation and social activities.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 years and older;
2. Diagnosis of unipolar major depression;
3. Montgomery Asberg Depression Rating Scale score ≥ 18;
4. Capacity to provide written consent for both research assessment and treatment;
5. Command of English sufficient to participate in assessments and talking therapy.

Exclusion Criteria:

1. Moderately severe to severe dementia (MMSE score < 20);
2. Greater than mild to moderate aphasia (NIH Stroke Scale: Best Language > 1);
3. Expectation to be discharged to a nursing home;
4. Psychotic depression;
5. Suicidal intent or plan.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Depression | 12 months
  This research study involves testing a modified form of problem-solving therapy called Ecosystem Focused Therapy (EFT) in reducing depression in older adult stroke survivors.

CONTACTS AND LOCATIONS:
Overall Officials: George S. Alexopoulos, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - New York Presbyterian Hospital, New York, New York
  - Burke Rehabilitation Hospital, White Plains, New York
  - Institute of Geriatric Psychiatry, White Plains, New York

IPD SHARING:
Plan to Share IPD: No